CLINICAL TRIAL: NCT07214415
Title: Evaluating the Effects of Hyperbaric Oxygen Therapy on Cognitive Function, Mental Health, and Quality of Life in Veterans
Brief Title: Veterans' Cognitive Function, Mental Health, and Quality of Life After Hyperbaric Oxygen Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Summit Hyperbarics and Wellness (Other)
Responsible Party: Principal Investigator, Steve Wyman, Medical Director, Summit Hyperbarics and Wellness
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBOT-VET-2025-001; 20253309 (Other: WIRB)
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: TBI Traumatic Brain Injury; PTSD - Post Traumatic Stress Disorder; Post Concussive Syndrome
MeSH Terms: conditions — Brain Injuries, Traumatic; Combat Disorders; Post-Concussion Syndrome | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HBOT Intervention Group (Experimental)
  Interventions: Drug: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Drug: Hyperbaric Oxygen Therapy — Each HBOT session is scheduled for approximately 95 minutes. The session will begin with a descent of up to 15 minutes (longer if needed for comfort/safety) to a pressure of 2.0 ATA, followed by 30 minutes of breathing 100% oxygen. At the midpoint, there will be a 5-minute air break from oxygen, after which subjects resume breathing 100% oxygen for another 30 minutes. Finally, the session will conclude with an ascent of up to 15 minutes (longer if needed for comfort/safety) back to 1.0 ATA.
  All sessions are delivered under direct medical supervision with standardized safety protocols. Once approved after medical and behavioral screening, participants complete a battery of cognitive, mental health, and quality of life assessments at baseline (pre-) and after completing the therapy (post-). This arm is distinct from any sham or control interventions because all participants receive the active HBOT treatment.

SUMMARY:
The purpose of this study is to evaluate how hyperbaric oxygen therapy (HBOT) may affect cognitive functioning, post-traumatic stress disorder (PTSD), depression, anxiety, and overall quality of life in veterans.

1. Does Hyperbaric Oxygen Therapy improve cognitive functioning, psychological well-being, and quality of life among veterans, as measured by pre-and post-treatment scores?
2. To what extent does Hyperbaric Oxygen Therapy improve cognitive functioning, psychological well-being, and qualify of life among veterans, after controlling for demographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Veteran status
3. Clinically diagnosed with a mTBI, PTSD, Anxiety, or Depression disorder by meeting the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, and by a qualified and trained professional.
4. The subject is willing and able to read, understand, and sign an informed consent. Additionally, the subject has clear consciousness and the ability to express self-feelings independently.
5. Exposed to at least one trauma-focused therapy or evidence-based psychotherapeutic treatment, such as prolonged exposure therapy, EMDR, or CBT, to name a few.
6. Completed cognitive and psychological measurements.
7. Clinical diagnoses cause significant impairment in social or occupational functioning or some other functional capacity.
8. Sexually active female participants of childbearing potential and sexually active male participants with female partners of childbearing potential must agree to use an acceptable method of contraception for the duration of the study and for 30 days following the final HBOT session.
9. Stability on any current psychoactive medications (antidepressants, anti-anxiety medications, antipsychotics, stimulants, and mood stabilizers).

Exclusion Criteria:

1. Untreated pneumothorax
2. History of spontaneous pneumothorax
3. Severe sinus infection
4. Upper respiratory infection
5. Asymptomatic pulmonary lesions on chest x-ray
6. Uncontrollable high fever (greater than 39C)
7. History of chest or ear surgery
8. Congenital spherocytosis
9. Any anemia or blood disorder
10. Any convulsive disorder
11. History of optic neuritis or sudden blindness
12. Middle ear infection
13. Diabetes mellitus (insulin therapy)
14. The subject is pregnant or lactating
15. Nicotine use/substance use/addiction
16. Acute Hypoglycemia
17. Diagnosed Chronic Obstructive Pulmonary Disease (COPD) and Emphysema
18. Presenting with symptoms of cough, congestion, vomiting, diarrhea, or open wounds.
19. Active malignancy
20. Current manic, delusional, or psychotic episodes
21. Serious/current suicidal ideations
22. Severe or unstable physical disorders or major cognitive deficits
23. Inability to attend scheduled clinic visits or comply with study protocols.
24. Treated with HBOT for any reason prior to study enrollment.
25. Non-English speakers
26. History of retinal repair, including laser photocoagulation or retinal detachment surgery.
27. History of middle ear surgery, including tympanoplasty, mastoidectomy, or pressure equalization tube placement.
28. Age greater than 75 years.
29. Use of any of the following medications during the study period: Anti-metabolites (e.g., methotrexate, azathioprine); Chemotherapuetic agents (e.g., cyclophosphamide, cisplatin); Mafenide acetate e.g., Sulfamylon); Disulfiram (e.g, Antabuse); Peripheral vasodilators known to interact with oxygen exposure (e.g., nitroglycerin); and Antibacterial drugs with known HBOT interaction risks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | From baseline assessment prior to first HBOT session to immediately after completion of final HBOT session
  Self-report questionnaire to assess symptoms of PTSD
NeuroTrax | From baseline assessment prior to first HBOT session to immediately after completion of final HBOT session.
  A computerized cognitive test to measure various cognitive functions, including memory, executive functioning, visual-spatial perception, verbal function, attention, information processing speed, and motor skills.
Patient Health Questionnaire-9 (PHQ-9) | From baseline assessment prior to first HBOT session to immediately after completion of final HBOT session
  Self-report questionnaire to assess depression severity
Generalized Anxiety Disorder 7-item scale (GAD-7) | From baseline assessment prior to first HBOT session to immediately after completion of final HBOT session
  Self-report questionnaire to measure anxiety severity
World Health Organization Quality of Life (WHOQOL-BREF) | From baseline assessment prior to first HBOT session to immediately after completion of final HBOT session
  Self-report questionnaire to rate a person's perception of his/her position in their life in the context of physical, psychological, level of independence, social relationships, environment, and spirituality/religion/personal belief domains and facets

CONTACTS AND LOCATIONS:
Overall Officials: Steven Wyman, MD, Principal Investigator — Summit Hyperbarics and Wellness
Locations (1):
- Summit Hyperbarics and Wellness, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: Undecided